CLINICAL TRIAL: NCT07358988
Title: A Multicenter Phase I Clinical Study of CD19-Targeted CAR-NK Cell Therapy for Moderate to Severe Active Systemic Lupus Erythematosus in China
Brief Title: KN5501 Cell Injection for Refractory SLE(CLEAR)
Acronym: CLEAR
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Ruitherapeutics Co., LTD (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: RUI-KN5501-SIL01
Record Dates: First submitted 2026-01-01; First posted 2026-01-22 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Systemic Lupus Erthematosus (SLE)

STUDY DESIGN:
Intervention Model Description: Part 1(SAD)：establish Maximum Tolerated Dose for single-dose setting, and dosing regimen for MAD; Part 2(MAD and expansion): establish Recommended Phase 2 Dose(RP2D)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- KN5501 cell injection (Experimental): inter-patient dose escalation arm with six dose levels for single-dose setting and 2-4 dose levels for multiple-dose setting
  Interventions: Drug: KN5501 cell injection

INTERVENTIONS:
Drug: KN5501 cell injection — In Part 1(SAD), six different doses will be explored to establish maximum tolerated dose for single-dose setting; In part 2(MAD and expansion), about 2-4 multiple-dose dosing regimen will be explored, and cohorts of 1-2 dosing regimen will be selected to expand.

SUMMARY:
The goal of this clinical trial is to learn about the safety, pharmacokinetics and pharmacodynamics profile of KN5501 cell injection in adults with systemic lupus erythematosus(SLE). It will also learn if KN5501 cell injection works to treat refractory SLE. The main questions it aims to answer are:

1. Is KN5501 cell injection safe in adults with SLE? And the maximum tolerated dose?
2. Does KN5501 cell injection lower the disease activity of SLE in adults with refractory SLE？

Participants will:

Receive one or multiple (3 to 5 times) intravenous infusion of KN5501 cell injection at inpatient ward after lymphodepletion.

Visit the clinic at predefined frequency (from 1 week interval to 12-16 weeks' interval) for checkups and tests.

ELIGIBILITY:
Inclusion Criteria:

* 1. Aged 18~70(including thresholds) when obtaining informed consent;
* 2. Body weight > 40.0 kg at screening;
* 3. Refractory SLE patients with moderate to severe activity;
* 4. CBC meeting predefined requirements at screening, including ANC ≥ 1.5×10^9/L, Hb ≥ 80g/L, and PLT ≥ 50×10^9/L(Not applicable, if it is ITP due to active SLE disease which is judged by investigator);
* 5. Adequate liver, kidney, lung and ;heart function at screening;
* 6. The date of last supportive therapy of hemopoietic growth factor(including EPO, G-CSF, GM-CSF and TPO, etc.)should be at least 2 weeks before screening visit, the last date of PLT infusion should be at least one week before screening visit, and the last date of RBC infusion should be at least 2 weeks before screening visit;
* 7. The number of CD19+ B cells in peripheral blood > 5 cells per microliter at screening;
* 8. Negative serum pregnancy test for WOCBPs at screening. Male or Female trial participants of child bearing potential should utilize efficient contraceptive measures from ICF signing until at least one year since the last dose, and promise not to donate ovums or sperms until at least one year since the last dose.

Exclusion Criteria:

* 1. Hypersensitive or allergic to any components of KN5501(e.g. DEXTRAN 40) or other trial interventions including fludarabine, cyclophosphamide, and tocilizumab, or having ever experienced severe anaphylaxis;
* 2. Severe lupus nephritis patients, defined as proteinuria ≥3.5g/24h or a history of renal replacement therapy. Or high risk of progressive LN disease which will probably require induced intensive treatment;
* 3. CNS affected, including but not limited to lupus encephalopathy, seizure, strock(ischemic or hemorrhagic), dementia, cerebellar disease, organic brain syndrome, encephalitis, CNS vasculitis, or mental disease;
* 4. Severe lung disease, e.g. pulmonary hypertension ≥ grade 3(WHO), or requiring mask oxygen therapy or ventilator-assisted breathing(non-invasive or invasive) ;
* 5. Unstable cardiovascular system, e.g. myocardial infarction within 6 months before screening, unstable angina within 3 months before screening, uncontrolled and clinically significant ventricular arrhythmia(including ventricular tachycardia, ventricular fibrillation, or TdP), second-degree atrioventricular block of Mobitz type II or third-degree atrioventricular block, congestive heart failure with New York Heart Association class ≥ 3; poorly controlled hypertension (SBP > 160 mmHg and/or DBP > 100 mmHg), or accompanied by hypertensive crisis or hypertensive encephalopathy;
* 6. Malignancy within 5 years before screening, excluding tumors with negligible risk of metastasis or death that are curable, such as radically treated non-melanoma skin cancer, localized prostate cancer, biopsy-confirmed cervical carcinoma in situ or squamous intraepithelial lesions detected by cervical smears, and completely resected ductal carcinoma in situ of the breast;
* 7. Severe infections requiring intravenous anti-infection treatment within 14 days before planned lymphodepletion, however preventive therapy is permitted;
* 8. Active or latent tuberculosis at screening;
* 9. HBV or HCV infection at screening. If positve HBsAg and/or HBcAb, HBV-DNA should be tested to confirm. If positive HCV-Ab, HCV-RNA should be tested to confirm;
* 10. Active HIV infection history, or positive serum HIV antigen or antibody test, or positive antibody test for Treponema Pallidum at screening.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 36 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2027-07 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
Dose Limiting Toxicity | from the first dose to 2 weeks (SAD) or 4 weeks (MAD)
Number of participants with adverse events | from enrollment to the last assessment at 52 weeks
  Number of participants with adverse events(including abnormal physical examinations(PE), abnormal vital signs, abnormal laboratory test results and abnormal 12-ECG readings

SECONDARY OUTCOMES:
Time to Peak Plasma Concentration (Tmax) | from the first dose to 4 weeks.
Peak Plasma Concentration (Cmax) | from the first dose to 4 weeks
Area under the plasma concentration versus time curve (AUC) | from the first dose to 4 weeks.
Duration of retention | from the first dose to 4 weeks
Number of CD19+ B cells per microlitre in peripheral blood (PD biomarker) | from enrollment to the last assessment at 52 weeks
Concentration of cytokines (IL-6, etc.) in peripheral blood (PD biomarker) | from enrollment to the last assessment at 52 weeks
Concentration of immunoglobulins (IgG, IgM, IgE and IgA) in peripheral blood (PD biomarker) | from enrollment to the last assessment at 52 weeks
Concentration of serum complements (PD biomarker) | from enrollment to the last assessment at 52 weeks
Number or percentage of B cell subsets in peripheral blood (PD biomarker) | from enrollment to the last assessment at 52 weeks
Response rate of DORIS 2021(The 2021 Definitions Of Remission In SLE) | from enrollment to the last assessment at 52 weeks
Response rate of LLDAS (Lupus Low Disease Activity Status) | from enrollment to the last assessment at 52 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Mengtao Li, Principal Investigator — Rheumatology Department, Peking Union Medical College Hospital
Locations (6):
- China (6):
  - Bengbu Medical College First Affiliated Hospital, Bengbu, Anhui
  - Peking Union Medical College Hospital, Beijing, Beijing Municipality
  - The First Affiliated Hospital of Henan University of Science and Technology, Luoyang, Henan
  - Union Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei
  - Jiangsu Provincial People's Hospital, Nanjing, Jiangsu
  - Changhai Hospital of Shanghai, Shanghai, Shanghai Municipality

IPD SHARING:
Plan to Share IPD: Yes
only IPD used in the results publication will be shared.